CLINICAL TRIAL: NCT00139958
Title: Prognosis After Acute Coronary Syndrome in HIV-infected Patients
Brief Title: Prognosis of Acute Coronary Syndrome in HIV-infected Patients
Status: Completed | Type: Observational
Sponsor: Saint Antoine University Hospital (Other)
Responsible Party: SAint Antoine University Hospital, Assistance publique Hôpitaux de Paris
Other Study IDs: PACS
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Heart Disease; HIV Infection
Keywords: Acute coronary syndrome; HIV infection; Prognosis; Coronary heart disease; Revascularization
MeSH Terms: conditions — Coronary Disease; HIV Infections; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lipids, CRP, glycemia, insulinemia
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Objectives: Evaluate differences for mortality, morbidity and the cardiovascular risk factors between HIV and non-HIV patients with an acute coronary syndromes (ACS) after a 3-years follow up.

DETAILED DESCRIPTION:
Background: There have been many cases of myocardial infarction reported in HIV-infected young adults treated with HAART. Little is known to date, concerning the outcome and prognostic factors of patients with acute coronary syndrome and HIV-infection.

Methods: Prospective cohort study to compare the evolution and prognosis between HIV and non-HIV patients with an ACS.

Duration of the study: Two years for including patients. Three years of follow-up 100 HIV-patients with ACS and 200 non-HIV patients with ACS will be included in the study. All patients will be included in the study from 30 Intensive Care Unit of Cardiology departments in France.

Results: To compare the incidence of total mortality, cardiovascular mortality (myocardial infarction, sudden death, cardiogenic shock, fatal stroke), morbidity (non fatal myocardial infarction, unstable angina, recurrence of ischemia, cardiac failure, non fatal stroke) and revascularization (percutaneous coronary intervention, coronary artery bypass graft surgery) during a 3-year follow-up between HIV and non-HIV patients with ACS. Univariate and multivariate analysis of predictive factors for cardiovascular events will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 year's old
* Man or woman HIV-infected for HIV 1 with or without highly active antiretroviral therapy
* Acute coronary syndromes (STEMI, NSTEMI and unstable angina)

Exclusion Criteria:

* Known atherosclerotic artery disease (MI, ACS, PCI, CABG, coronary stenosis, stroke, peripheral arteriopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAtients with de novo acute coronary syndromes age > 18years old.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2003-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the rate of Major Adverse Cardiac and Cerebrovascular Events between HIV+ and HIV- after a first episode of ACS after a 3-years follow up. | 36 months

SECONDARY OUTCOMES:
Clinical, angiographic characteristics at baseline and comparison between HIV+ and HIV- | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Cohen, MD, PhD, Study Chair — Saint Antoine University Hospital
Locations (1):
- Cardiology department, Paris, France

REFERENCES:
- [Derived] Robert R, Cottin Y, Potard V, Mary-Krause M, Lang S, Teiger E, Collet JP, Chauvet-Droit M, Ederhy S, Soulat-Dufour L, Ancedy Y, Adavane-Scheuble S, Nhan P, Steg PG, Funck-Brentano C, Costagliola D, Cohen A, Boccara F; on behalf the PACS-HIV Investigators. Coronary Angiographic Features and Major Adverse Cardiac or Cerebrovascular Events in People Living With Human Immunodeficiency Virus Presenting With Acute Coronary Syndrome. Circ Cardiovasc Interv. 2022 Jun;15(6):e011945. doi: 10.1161/CIRCINTERVENTIONS.122.011945. Epub 2022 May 10. No abstract available. PMID 35535605
- [Derived] Boccara F, Mary-Krause M, Potard V, Teiger E, Lang S, Hammoudi N, Chauvet M, Ederhy S, Dufour-Soulat L, Ancedy Y, Nhan P, Adavane S, Steg PG, Funck-Brentano C, Costagliola D, Cohen A; PACS-HIV (Prognosis of Acute Coronary Syndrome in HIV-Infected Patients) Investigators dagger. HIV Infection and Long-Term Residual Cardiovascular Risk After Acute Coronary Syndrome. J Am Heart Assoc. 2020 Sep;9(17):e017578. doi: 10.1161/JAHA.119.017578. Epub 2020 Aug 26. PMID 32844734